CLINICAL TRIAL: NCT03910374
Title: Role of Leukocyte- and Platelet-Rich Fibrin Membranes in Endoscopic Endonasal Skull Base Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Laura Van Gerven, Clinical professor, Doctor, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: s61636
Record Dates: First submitted 2019-03-20; First posted 2019-04-10 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Cranial Sutures; Closure
Keywords: L-PRF; fibrin sealants; endoscopic endonasal skull base reconstruction

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Participant
Masking Description: Participants stay masked during the trial, care provider and investigators are unblinded at the surgical procedure and from thereon
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classical Treatment (Placebo Comparator): In this arm, dural closure will be performed with the classical fibrine sealants.
  Interventions: Procedure: Dural closure
- L-PRF (Active Comparator): In this arm, dural closure will be performed with the autologous L-PRF
  Interventions: Procedure: Dural closure

INTERVENTIONS:
Procedure: Dural closure — Evaluation of the safety and effectiveness of autologous blood-derived products (L-PRF and fibrinogen) compared to the fibrin sealants as an adjunct for dural repair

SUMMARY:
Prospective investigation of the effectivity of L-PRF membranes for skull base reconstruction after endoscopic endonasal skull base surgery (transsphenoidal) versus classical closure techniques.

DETAILED DESCRIPTION:
The investigators want to demonstrate in a prospective, randomized trial including 220 patients undergoing endoscopic endonasal skull base surgery that the use of L-PRF is non-inferior to classical fibrin sealants.

Approximately 220 patients undergoing cranial surgery will be enrolled in this randomized, controlled, single-blinded multicenter study to evaluate the safety and effectiveness of autologous blood-derived products (L-PRF and fibrinogen) compared to the fibrin sealants as an adjunct for dural repair.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lesions of the sellar/parasellar region
* Age > 18 and < 70 years
* Written informed consent
* Willingness to adhere to visit schedules

Exclusion Criteria:

* Age < 18 and > 70 years
* Any underlying rhinological condition like nasal polyps, which may interfere with the obtained results
* Any disorder which might compromise the ability of a patient to give truly informed consent for participation in this study
* Enrollment in other investigational drug trial(s)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
To compare the prevalence of CSF-leaks after L-PRF closure and after the classical closure techniques for sellar defects to demonstrate non-inferiority | 4 years
  The primary aim of this study is identifying the role of L-PRF in the endoscopic endonasal closure of skull base defects. More specific, we want to demonstrate in a prospective, randomized trial that the use of L-PRF is non-inferior to classical closure techniques regarding prevalence of CSF-leaks The number of patients with a CSF-leak will be compared between both treatment groups.
Cost-effectiveness evaluation based on the effectiveness and the costs of L-PRF versus the current golden standard (Tachosil and Tisseel). | 4 years
  Cost-effectiveness evaluation: compare the costs and the effectiveness of L-PRF versus commercial fibrin sealants.

SECONDARY OUTCOMES:
To identify potential risk for closure-failures based on the size of the lesion | 4 years
  The potential risk for closure-failure (evaluated by the prevalence of CSF-leaks) based size of lesion ( evaluated by Wilson-Hardy classification) will be measured.
To evaluate if the pathology is a potential risk factor for closure-failures | 4 years
  The potential risk for closure-failure (evaluated by the prevalence of CSF-leaks) based on the pathology will be evaluated.
To evaluate if the age of the patient is a potential risk factor for closure-failures | 4 years
  The potential risk for closure-failure (evaluated by the prevalence of CSF-leaks) based on the age of the patients will be measured.
Evaluate the effect of L-PRF versus the current golden standard (Tachosil and Tisseel) on post-operative symptoms based on a visual analogue scale | 4 years
  Rhinological symptoms as well as quality of life before and after surgery will be assesed using a visual analogue scale. The symptoms will be scored on a horizontal line of 10 cm, where 0 cm equals "no symptoms" and 10 cm equals "very severe symptoms".
Evaluate the effect of L-PRF versus the current golden standard (Tachosil and Tisseel) on post-operative symptoms based on the SNOT-22 | 4 years
  Rhinological symptoms as well as quality of life before and after surgery will be assesed using a SNOT-22. The symptoms will be scored between 0 and 5 where 0 equals "no symptoms" and 5 equals "very severe symptoms".
Evaluate the effect of L-PRF versus the current golden standard (Tachosil and Tisseel) on post-operative symptoms based on the skull base questionnaire | 4 years
  Rhinological symptoms as well as quality of life before and after surgery will be assesed using the skull base questionnaire.
Evaluate the effect of L-PRF versus the current golden standard (Tachosil and Tisseel) on post-operative symptoms based on the EQ-5D | 4 years
  Rhinological symptoms as well as quality of life before and after surgery will be assesed using the EQ-5D
Evaluate the potential interference of the L-PRF membranes with post-operative imaging by comparing the tumor residue evaluation 3 months and 1 year after surgery | 4 years
  potential interference of the L-PRF membranes with post-operative imaging (MRI) will be evaluated. 3 months after surgery, when the L-PRF membrane is still visible, the MRI images will be evaluated to see if there is tumor residue present or not. After 1 year the presence of tumor residue will be reevaluated. The outcomes will be compared between both evaluation timepoints to asses if L-PRF has interference with the imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Van Gerven, prof, Principal Investigator — UZ Leuven
Locations (3):
- Belgium (2):
  - AZ Sint-Jan, Bruges
  - UZ Leuven, Leuven
- Fundació Clínic Per A La Recerca Biomèdica, Barcelona, Spain

REFERENCES:
- [Derived] Coucke B, Van Hoylandt A, Jorissen M, Meulemans J, Decramer T, van Loon J, Vander Poorten V, Theys T, Van Gerven L. Leukocyte- and platelet-rich fibrin in endoscopic endonasal skull base reconstruction: study protocol for a multicenter prospective, parallel-group, single-blinded randomized controlled non-inferiority trial. Trials. 2023 Jul 31;24(1):488. doi: 10.1186/s13063-023-07492-w. PMID 37525278